CLINICAL TRIAL: NCT07177794
Title: Toripalimab Combined With Capecitabine as Maintenance Therapy After Definitive Chemoradiotherapy for Esophageal Squamous Cell Carcinoma: a Multicenter, Randomized Controlled, Phase III Trial (EC-CRT-008)
Brief Title: Consolidation of Toripalimab and Capecitabine After Chemoradiotherapy in ESCC
Acronym: EC-CRT-008
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Collaborators: First Affiliated Hospital, Sun Yat-Sen University (Other); Fifth Affiliated Hospital, Sun Yat-Sen University (Other); Zhongshan People's Hospital, Guangdong, China (Other)
Responsible Party: Principal Investigator, Mian XI, Professor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B2025-404-01
Record Dates: First submitted 2025-09-10; First posted 2025-09-17 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Esophageal Cancer; Chemoradiotherapy
Keywords: Esophageal squamous cell carcinoma; definitive chemoradiotherapy; maintenance therapy; Toripalimab
MeSH Terms: conditions — Esophageal Neoplasms; Esophageal Squamous Cell Carcinoma | interventions — toripalimab; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A (Experimental): Patients will receive toripalimab combined with metronomic capecitabine, with a maximum treatment duration of one year (toripalimab 240 mg, IV drip, Q3W, for 16 cycles; capecitabine 500 mg, twice daily, orally).
  Interventions: Drug: toripalimab; Drug: capecitabine
- Arm B (No Intervention): Patients will undergo conventional observation and follow-up.

INTERVENTIONS:
Drug: toripalimab — Patients will receive toripalimab with a maximum treatment duration of one year (240 mg, IV drip, Q3W, for 16 cycles).
  Other Names: JS001
  Arms: Arm A
Drug: capecitabine — Patients will receive metronomic capecitabine, with a maximum treatment duration of one year (500 mg, twice daily, orally).
  Other Names: Xeloda
  Arms: Arm A

SUMMARY:
Definitive chemoradiotherapy (CRT) is the standard treatment for locally advanced unresectable esophageal cancer, but its efficacy remains unsatisfactory. More importantly, there is a lack of effective consolidation treatment after CRT, resulting in a high recurrence rate. Our previous prospective phase II trial (EC-CRT-001) demonstrated that the addition of toripalimab to definitive CRT improved the complete response rate in patients with locally advanced esophageal squamous cell carcinoma (ESCC), showing potential for enhanced long-term survival with a manageable safety profile. Nevertheless, the risk of recurrence requires further reduction. Metronomic capecitabine chemotherapy can modulate the tumor immune microenvironment and may synergize with PD-1 antibodies to enhance antitumor efficacy, potentially further prolonging survival in ESCC. Based on current research advances and our preliminary findings, this randomized, controlled, multicenter, phase III clinical trial aims to evaluate the efficacy and safety of toripalimab combined with capecitabine as maintenance therapy for patients with locally advanced ESCC who have not progressed after definitive CRT.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed squamous cell carcinoma of the esophagus;
2. Locally advanced esophageal cancer classified as stage I-IVA (inoperable or patient declined surgery) or stage IVB thoracic esophageal cancer with supraclavicular lymph node metastasis only (AJCC 8th edition) prior to treatment;
3. Completion of definitive concurrent chemoradiotherapy without disease progression; radiotherapy dose of 50-50.4 Gy using conventional fractionation and IMRT technique; concurrent platinum- or taxane-based doublet chemotherapy during radiotherapy; ≤4 cycles of induction chemotherapy allowed prior to radiotherapy; PD-1/PD-L1 antibody therapy permitted during induction chemotherapy and radiotherapy; no adjuvant therapy received;
4. Enrollment window: within 1-42 days after completion of chemoradiotherapy;
5. Age 18-75 years;
6. Estimated life expectancy >6 months;
7. Eastern Cooperative Oncology Group performance status ≤ 2;
8. The function of important organs meets the following requirements: a. white blood cell count (WBC) ≥3.5×109/L, absolute neutrophil count (ANC) ≥1.5×109/L; b. platelets ≥75×109/L; c. hemoglobin ≥9g/dL; d. serum albumin ≥2.8g/dL; e. total bilirubin ≤1.5×ULN, ALT, AST and/or AKP ≤2.5×ULN; f. serum creatinine ≤1.5×ULN or creatinine clearance rate >60 mL/min;
9. Ability to understand the trial details and has provided written informed consent.

Exclusion Criteria:

1. Patients who have received antitumor therapy (including adjuvant chemotherapy, surgery, immunotherapy, targeted therapy, etc.) after completion of chemoradiotherapy;
2. Stage IVb patients with metastasis to solid organs (e.g., liver, bone, lung, brain, adrenal gland, peritoneum, etc.) at initial diagnosis;
3. Known or suspected allergy to the investigational drug(s) or any agent related to the trial regimen;
4. Presence of esophageal fistula and/or esophageal hemorrhage prior to enrollment;
5. Disease progression after chemoradiotherapy;
6. ≥Grade 2 radiation pneumonitis prior to enrollment;
7. History of ≥ Grade 3 immune-related adverse events prior to enrollment;
8. Prior treatment with targeted drugs;
9. History of other malignant tumors besides esophageal cancer, except for non-melanoma skin cancer, carcinoma in situ of the cervix, papillary thyroid carcinoma, or cured early-stage prostate cancer;
10. Patients with severe cardiac, pulmonary, hepatic, or renal dysfunction, hematopoietic system diseases, cachexia, or other conditions that make them unfit for chemotherapy;
11. Female patients who are pregnant or breastfeeding;
12. Inability to provide informed consent due to psychological, familial, social, or other factors;
13. Presence of CTC grade ≥2 peripheral neuropathy;
14. Patients with a history of diabetes for more than 10 years and poorly controlled blood glucose levels;
15. History of autoimmune disease or autoimmune disorders (e.g., colitis, systemic lupus erythematosus, rheumatoid arthritis, uveitis, hypophysitis, hyperthyroidism; not limited to these diseases or syndromes), immunodeficiency history, including HIV positivity, or other acquired/congenital immunodeficiency disorders, or history of organ transplantation or allogeneic bone marrow transplantation;
16. History of interstitial lung disease or non-infectious pneumonia;
17. Active hepatitis B (HBV DNA ≥2000 IU/mL or 10⁴ copies/mL) or hepatitis C (HCV antibody positive with HCV-RNA above the lower limit of detection);
18. Any unstable condition that may jeopardize patient safety or compliance.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 242 (Estimated)
Dates: Start 2025-09-20 (Estimated); Primary Completion 2028-05-31 (Estimated); Study Completion 2030-05-31 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival | From date of enrollment until the date of death from any cause or the date of first documented disease progression whichever came first, assessed up to 36 months
  Three-year follow-up from the date of enrollment to the date of disease progression or last follow-up

SECONDARY OUTCOMES:
Overall survival | From date of enrollment until the date of death from any cause or the date of last follow-up, whichever came first, assessed up to 36 months
  Three-year follow-up from the enrollment to the date of death from any cause or date of lost follow-up
Clinical complete response | 14-16 weeks after the completion of radiotherapy
  Tumor response was evaluated 14-16 weeks after the completion of radiotherapy based on CT or PET-CT scans, and endoscopy with biopsies.
Treatment-related adverse events | From date of enrollment to the date of last follow-up, assessed up to 36 months.
  Incidence of treatment-related adverse events as assessed by CTCAE v4.0.

OTHER OUTCOMES:
Correlation between immune signature and overall survival | From date of enrollment to the date of last follow-up, assessed up to 36 months.
  The correlation between pretreatment immune signature (PD-L1, CD8, CTLA-4, CD56, and CD68) by mIHC and overall survival.
Correlation between dynamic change of ctDNA and overall survival | From date of enrollment to the date of last follow-up, assessed up to 36 months.
  The correlation between dynamic change of ctDNA during treatment and survival outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Mian Xi, MD, Principal Investigator — Sun Yat-sen University
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Zhu Y, Wen J, Li Q, Chen B, Zhao L, Liu S, Yang Y, Wang S, Lv Y, Li J, Zhang L, Hu Y, Liu M, Xi M. Toripalimab combined with definitive chemoradiotherapy in locally advanced oesophageal squamous cell carcinoma (EC-CRT-001): a single-arm, phase 2 trial. Lancet Oncol. 2023 Apr;24(4):371-382. doi: 10.1016/S1470-2045(23)00060-8. PMID 36990609
- [Result] Bando H, Kumagai S, Kotani D, Mishima S, Irie T, Itahashi K, Tanaka Y, Habu T, Fukaya S, Kondo M, Tsushima T, Hara H, Kadowaki S, Kato K, Chin K, Yamaguchi K, Kageyama SI, Hojo H, Nakamura M, Tachibana H, Wakabayashi M, Fukui M, Fuse N, Koyama S, Mano H, Nishikawa H, Shitara K, Yoshino T, Kojima T. Atezolizumab following definitive chemoradiotherapy in patients with unresectable locally advanced esophageal squamous cell carcinoma - a multicenter phase 2 trial (EPOC1802). Nat Cancer. 2025 Mar;6(3):445-459. doi: 10.1038/s43018-025-00918-1. Epub 2025 Feb 19. PMID 39972105
- [Result] Jia R, Shan T, Zheng A, Zhang Y, Lu P, Zhang G, Wang F, Xu Z, Zheng G, Tang D, Zhang W, Li W, Li R, Guo Y, Liu L, Luo X, Zheng Y, Chang Z, Wang Q, Wang X, Yuan X, Kong G, Li S, Yang R, Zhou D, Ren J, Yin W, Li J, Zhang J, Wang Z, Sheng M, Xu B, Li L, Liu X, Lu Z, Wan L, Zhou F, Gao S. Capecitabine or Capecitabine Plus Oxaliplatin Versus Fluorouracil Plus Cisplatin in Definitive Concurrent Chemoradiotherapy for Locally Advanced Esophageal Squamous Cell Carcinoma (CRTCOESC): A Multicenter, Randomized, Open-Label, Phase 3 Trial. J Clin Oncol. 2024 Jul 10;42(20):2436-2445. doi: 10.1200/JCO.23.02009. Epub 2024 May 6. PMID 38710003